CLINICAL TRIAL: NCT05531500
Title: Patient Reported Outcomes Following Interventional Procedures in Pelvic Pain
Acronym: pelvicpain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Medhat Farghaly, Assistant lecturer of anesthesia , Intensive care and pain medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pelvic pain outcome
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Pudendal Neuralgia
Keywords: Pelvic pain
MeSH Terms: conditions — Pudendal Neuralgia; Pelvic Pain | interventions — Injections

STUDY DESIGN:
Intervention Model Description: parallel groups of different intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection (Other): Injection of local anesthetic and steroid to the diseased nerve
  Interventions: Drug: Injection
- Radiofrequency (Other): Application of radiofrequency to the diseased nerve
  Interventions: Device: Radiofrequency

INTERVENTIONS:
Drug: Injection — Injection of local anesthetic + steroids
  Arms: Injection
Device: Radiofrequency — Application of radiofrequency on the diseased nerve
  Arms: Radiofrequency

SUMMARY:
The investigators aim from this study, to determine the safety and efficacy of pulsed radiofrequency in the management of pudendal neuralgia, compared to current a standard intervention, which is corticosteroid injection for PN, as part of multidisciplinary pain management.

DETAILED DESCRIPTION:
The aim of this study is toillustrate whether pulsed radiofrequency treatment is safe and effective intreating the chronic perineal pain associated with PN or pudendal nerve compression; and whether it can be used as an integral part of its multidisciplinary managementBased on literature, the prevalence of Chronic Pelvic Pain (CPP) in general population ranges between 5.7% and 26.6%(Ahangari, 2014). There are many countries and regions with no published data in the field of CPP (Ahangari, 2014). CPP is a great burden to the patients and the healthcare systems (Latthe et al., 2006). About £154 million was the estimated cost of treatment for the women who suffer from CPP per year (Cheong and William Stones, 2006). CPP affects one's movement and their posture due to the secondary hyperalgesia in the pelvic muscles leading to diminished proprioception. About 50%- 70% of women with CPP have limitation on their daily activity(Ahangari, 2014). PN occurs in men, but the incidence/prevalence is not well studied. The principle therapy for chronic neuropathic pain is to eliminate the underlying causes of the pain (Belgrade, 2003), for PN this may involve surgical decompression. Pharmacotherapy and physiotherapy are two different options for treatment of neuropathic pain but they each come with limitations and drawbacks. Different techniques for pudendal nerve block have been described for managing PN but they have complications that may be serious such, vascular injury or intravascular injection with toxicity. The indication of surgery is in patients with failure of conservative treatment or other PNB techniques / modalities and includes decompression or neuromodulation.

Type of the study: A retrospective randomized controlled study Study Setting: University college London hospital

Sample Size Calculation:

Sample size calculation was carried out using G*Power 3 software (Faul et al., 2007). A calculated minimum sample of the cases is 60 patients, 30 in each group.

Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

Total number of the cases is 60 patients, 30 in each group.

Intervention(s):

1. Informed written consent: - A copy of the signed Informed Consent form will be given to the participant.

   The original signed form will be retained at the study site and a copy placed in the medical notes.
2. The patient is placed in the prone position
3. The ischial spine is then located using fluoroscopic X ray.
4. Aseptic cleaning of the skin in the target area
5. Patient will randomly be allocated to the control group receiving steroid and local anaesthetic injection or treatment group receiving pulsed radiofrequency treatment and local anaesthetic. Randomisation will be performed using sealed envelopes. I. Local anaesthetic and corticosteroid injection (control group)

   ▪ Under X-Ray guidance, the Needle (22G 5-10 cm insulated radiofrequency needle) is advanced perpendicular to the skin and placed transgluteally, directly avoiding the adjacent sciatic nerve at either the extremity of the ischial spine between the sacrotuberous and sacrospinous ligaments.
   * Sensory Electrostimulationis used to identify the nerve. For the motor stimulation, a unilateral contraction of the anal sphincter indicates that the inferior anal nerve had been stimulated while for the sensory stimulation, a sensation of tingling or numbness in the perineal region may be felt by the patient.
   * Contrast injected to avoid intravascular injection. A blinded operator sets the radiofrequency machine for a timer alert at five minutes.
   * After confirming the exact location of the needle tip, 4 mL of 1% lidocaine and 3.3 of dexamethasone in 1 mL are injected. II. Pulsed radiofrequency (Treatment/intervention group)
   * Needle is placed using the same technique as above and contrast medium is injected.
   * Lesion: - Radiofrequency current will be applied for 5 minutes, 120 ms, at 2 Hz, with maximum tissue temperature increased to 42°C. (usually not felt by the patient)
   * 4 mL of 1% lidocaine and 1 mL of NaCl .9% are injected.
6. Post procedure instructions:- ▪ Standard post procedure monitoring for 1 hour in theatre recovery, including treatment of nausea/vomiting and localized pain with standard intravenous/oral medication.

   * Immediate adverse events reporting.
   * Standard hospital post procedure instructions

Research outcome measures:

1. Primary Endpoint:

   Reduction in at least 1.5 point pain as measured by Numerical Rating Scale Secondary Endpoint A. NRS at 0, 1 and 12 weeks B Quality of Life Assessment at baseline, week 1, week 6 and week 12 a. EDQ5-5L b. SF-12 c. Brief Pain Inventory d. Global response Assessment C. Mood assessment at baseline, week 6 and week 12

   a. Pain Catastrophising Questionnaire b. Beck Depression Inventory II c. Hamilton Anxiety Rating Scale d. Sexual function assessment (questionnaire) at baseline, weeks 6 and 12 e. Lower urinary tract symptom assessment at baseline, weeks 6 and 12 f. Bristol Female Lower Urinary Tract Symptoms (BFLUTS-SF) g Review of pain medication use at weeks 6, 12 compared to baseline. h. Assessment of all patients against Nantes criteria at baseline

   2.5-Data management and analysis (Details needed): Data collection. Telephone review - Week 1
   1. Telephone review in 1 week to assess for complication and side effcte profile.
   2. Global pelvic pain NRS scores over telephone.
   3. Adverse events reporting.

   b. Telephone review at 6 weeks and 12 weeks
   1. review pelvic pain
   2. Questionaires: global pelvic pain, QoL and function
   3. Medication review

   <!-- -->

   1. S - Study/Statistical design (e.g. randomised controlled trial, case control study, pilot study):
   2. Prospective
   3. Parallel group ( 2 different groups)
   4. No active Control
   5. Randomized
   6. Single blinded
   7. multicentric study (at UCLH center)

   Statistical methods:

   i. All data will be collected and cleaned by Excel program then will be analyzed with SPSS software (Statistical Package for the Social Sciences, version 16, SSPS Inc, and Chicago, USA). ii. Continuous parametric data between two groups, two sample T test will be used.

   iii. Continuous parametric data between more than 2 groups, ANOVA test will be used.

   iv. Descriptive statistics will be done in the form of mean and standard error (SE).

   v. Frequency of qualitative variables and Chi-square test will be done. vi. In Categorical data, Chi-squared test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain> 6 months

  * Patients aged > 18years
  * Patients with unilateral or bilateral regional pelvic pain withpudendal irritation diagnosed by a pain clinician and clinically indicated to undergo pudendal nerve block by a consultant experienced in the field.

Exclusion Criteria:

* Known concurrent neurological or neurodegenerative disease, including those with impaired neurotransmission e.g. myasthenia gravis, multiple sclerosis, spinal cord injury etc

  * Pelvic surgery is expected within 3 months
  * Breastfeeding or pregnant women
  * Known current pelvic/pelvic organ infection or malignancy (Red flags)
  * Concurrent radiotherapy treatment to pelvis
  * Allergy/sensitivity to lidocaine anaesthetic or/ and corticosteroids therapy
  * Contraindication to receive a Pudendal nerve block eg high risk of bleeding
  * Active psychiatric or mental conditions ▪ Other uncontrolled medical condition

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-09 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 6months 1 year after intervention
  Pain score value from 1 to 10 reported by each individual patient following inter vention

CONTACTS AND LOCATIONS:
Overall Officials: Medhat SA Farghaly, master, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://link.springer.com/article/10.1007/s11608-006-0064-2 — https://link.springer.com/article/10.1007/s11608-006-0064-2
- See also: https://connect.springerpub.com/content/sgrcl/5/3/97.abstract — https://connect.springerpub.com/content/sgrcl/5/3/97.abstract
- See also: https://journals.lww.com/anesthesia-analgesia/FullText/2013/12000/The_Effectiveness_of_Pudendal_Nerve_Block_Versus.21.aspx — https://journals.lww.com/anesthesia-analgesia/FullText/2013/12000/The_Effectiveness_of_Pudendal_Nerve_Block_Versus.21.aspx
- See also: https://www.diva-portal.org/smash/record.jsf?pid=diva2:770659 — https://www.diva-portal.org/smash/record.jsf?pid=diva2:770659
- See also: https://bmcpublichealth.biomedcentral.com/articles/10.1186/1471-2458-6-177 — https://bmcpublichealth.biomedcentral.com/articles/10.1186/1471-2458-6-177
- See also: https://books.google.com/books?hl=ar&lr=&id=FMU0AwAAQBAJ&oi=fnd&pg=PP1&dq=+Chestnut+D,+Polley+L,+TsenL,Wong+C,+eds.+Chestnut%E2%80%99s+obstetric+anesthesia:+Principles+and+practice.&ots=czX9TVymak&sig=AVjCTsd6bT3TEKhgQ5BoBIJZuXg — https://books.google.com/books?hl=ar&lr=&id=FMU0AwAAQBAJ&oi=fnd&pg=PP1&dq=+Chestnut+D,+Polley+L,+TsenL,Wong+C,+eds.+Chestnut%E2%80%99s+obstetric+anesthesia:+Principles+and+practice.&ots=czX9TVymak&sig=AVjCTsd6bT3TEKhgQ5BoBIJZuXg